CLINICAL TRIAL: NCT04361318
Title: Clinical Trial Evaluating Safety and Efficacy of Hydroxychloroquine and Nitazoxanide Combination as Adjuvant Therapy in Covid-19 Newly Diagnosed Egyptian Patients: A Tanta University Hope
Brief Title: Hydroxychloroquine and Nitazoxanide Combination Therapy for COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kamal Mohammed Okasha, Vice-President of Postgraduate Studies and Research Affairs, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCQ/NTZ
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Hydroxychloroquine; Nitazoxanide; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; nitazoxanide; Drug Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: a double blind randomized controlled parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine plus Nitazoxanide (Experimental): 200 mg of Hydroxychloroquine orally three times daily for 10 days plus 500 mg of Nitazoxanide orally twice daily for 6 days
  Interventions: Combination Product: Hydroxychloroquine plus Nitazoxanide
- Standard care (Active Comparator): Standard care delivered in the COVID-19 isolation hospitals.
  Interventions: Other: Standard care

INTERVENTIONS:
Combination Product: Hydroxychloroquine plus Nitazoxanide — Both hydroxychloroquine & nitazoxanide will be administered orally to participating patients
  Other Names: drug therapy
  Arms: Hydroxychloroquine plus Nitazoxanide
Other: Standard care — Oxygen administered via ventilator. In addition, antipyretic "paracetamol" may be added if necessary
  Arms: Standard care

SUMMARY:
In December 2019, a new infectious respiratory disease emerged in Wuhan, Hubei province, China. An initial cluster of infections was linked to Huanan seafood market, potentially due to animal contact. Subsequently, human-to-human transmission occurred and the disease, now termed coronavirus disease 19 (COVID-19) rapidly spread within China and all over the world. A novel coronavirus, SARS-coronavirus 2 (SARS-CoV-2), which is closely related to SARS-CoV, was detected in patients and is believed to be the etiologic agent of the new lung disease. The causative agent of the current COVID-19 pandemic, SARS-CoV-2, is a single stranded positive sense RNA virus that is closely related to severe acute respiratory syndrome coronavirus (SARS-CoV).

DETAILED DESCRIPTION:
Selected Drugs

Hydroxychloroquine (an analog of chloroquine) has been demonstrated to have an anti-SARS-CoV activity in vitro. Hydroxychloroquine clinical safety profile is better than that of chloroquine (during long-term use) and allows higher daily dose and has fewer concerns about drug-drug interactions. Hydroxychloroquine has long-term safety (600 mg/day for 12 to 18 months was safe). Hydroxychloroquine effectively inhibited both the entry, transport and the post-entry stages of SARS-CoV-2, similar to the chloroquine, and one study found Hydroxychloroquine to be a more potent agent than chloroquine in inhibiting SARS-CoV-2 in vitro. Hydroxychloroquine acts as a weak base that can change the pH of acidic intracellular organelles including endosomes/lysosomes, essential for the membrane fusion. Besides, the significant decrease in the production of pro-inflammatory markers and cytokines with Hydroxychloroquine has made this agent a successful disease modifying anti-inflammatory agent in the treatment of various autoimmune diseases. An additional issue to be considered in severely sick patients is cytokine storm associated with disease severity of SARS-CoV-2.

There are no currently available data from randomized clinical trials (RCTs) to inform clinical guidance on the use, dosing, or duration of Hydroxychloroquine for prophylaxis or treatment of SARS-CoV-2 infection. Although optimal dosing and duration of Hydroxychloroquine for treatment of COVID-19 are unknown, some U.S. clinicians have reported anecdotally different Hydroxychloroquine dosing such as 400 mg twice daily on day one, then daily for 5 days; 400 mg twice daily on day one, then 200 mg twice daily for 4 days; 600 mg twice daily on day one, then 400 mg daily on days 2-5. In a recent clinical trial, Hydroxychloroquine sulfate 200 mg, three times per day during ten days was used in patients with COVID-19.

Nitazoxanide is originally developed as an antiprotozoal agent and has a broad-spectrum antiviral activity undergoing development for the treatment of influenza and other viral respiratory infections. In addition to its antiviral activity, Nitazoxanide inhibits the production of pro-inflammatory cytokines TNF-α, IL-2, IL-4, IL-5, IL-6, IL-8 and IL-10 in peripheral blood mononuclear cells. Nitazoxanide could improve outcomes in patients infected with MERS-CoV by suppressing overproduction of pro-inflammatory cytokines, including IL-6. Nitazoxanide has been tested in clinical setting for the treatment of acute uncomplicated influenza, where the subjects received either 600 or 300 mg of Nitazoxanide or placebo orally twice daily for five days and were followed for 28 days. Subjects who received Nitazoxanide 600 mg twice daily experienced shorter times to alleviation of symptoms compared with subjects who received 300 mg Nitazoxanide twice daily, which in turn, was shorter than placebo.

According to the National Health Commission of the People's Republic of China, there is lack of effective antiviral therapy against COVID-19. Nearly all patients who suffered from COVID-19-associated pneumonia accepted oxygen therapy and WHO recommended extracorporeal membrane oxygenation (ECMO) to patients with refractory hypoxemia. Rescue treatment with convalescent plasma and immunoglobulin G are delivered to some critical cases according to their condition.

The rationale of the use of Hydoxychloroquine and Nitazoxanide combination for treatment of COVID-19 infected patients is based on the antiviral and anti-inflammatory activity of the selected drugs. Since the two drugs exhibit different modes of action, it would be of value in containing the viral infection through targeting different sites in the pathophysiology of the disease.

Diagnostic criteria

The viral research institution in China has conducted preliminary identification of the SARS-CoV-2 through the classical Koch's postulates and observing its morphology through electron microscopy. So far, the golden clinical diagnosis method of COVID-19 is nucleic acid detection in the nasal and throat swab sampling or other respiratory tract samplings by real-time PCR and further confirmation by next-generation sequencing.

Side effects of Hydroxychloroquine

* The most common adverse effects are mild nausea and occasional stomach cramps with mild diarrhea, reduced appetite and vomiting
* The most serious adverse effects are retinopathy and heart problems
* Long term use may cause liver toxicity Contraindications of Hydroxychloroquine
* Heart conditions, diabetes or psoriasis.
* The drug transfers into breast milk so should be used with care by pregnant or nursing women

Interactions of Hydroxychloroquine

* Antacids may decrease the absorption of Hydroxychloroquine.
* Both neostigmine and pyridostigmine antagonize the action of Hydroxychloroquine.
* There may be a link between Hydroxychloroquine and hemolytic anemia in those with glucose-6-phosphate dehydrogenase deficiency.
* Digoxin; concomitant administration with Hydroxychloroquine may result in increased serum digoxin levels.
* Insulin or antidiabetic drugs; concomitant administration with Hydroxychloroquine may enhance the effects of the hypoglycemic treatment.
* Hydroxychloroquine prolongs the QT interval and may increase the risk of inducing ventricular arrhythmias if used concurrently with other arrhythmogenic drugs.
* Mefloquine and other drugs that lower the convulsive threshold, when co-administered with Hydroxychloroquine, there may be an increased risk of convulsions.
* Concurrent use of Hydroxychloroquine with antiepileptics may impair the antiepileptic activity.
* Cyclosporin when used concomitantly with Hydroxychloroquine, an increased plasma cyclosporin level was reported.

Side effects of Nitazoxanide

The most common adverse effects are GIT as nausea and occasional stomach cramps with mild diarrhea, reduced appetite and vomiting. Nervous system side effects as headache, dizziness, somnolence, insomnia, tremor, and hypesthesia have been reported in less than 1% of the patients.

Contraindications of Nitazoxanide

There are no data on the excretion of Nitazoxanide into human milk. The manufacturer recommends that caution be used when administering Nitazoxanide to nursing women.

Tizoxanide (the active metabolite of Nitazoxanide) is highly bound to plasma protein (> 99.9%). Therefore, it is necessary to monitor for adverse reactions when administering Nitazoxanide concurrently with other highly plasma protein-bound drugs with narrow therapeutic indices, as competition for binding sites may occur (e.g., warfarin).

Warning

Nitazoxanide should be used with caution in patients with significant renal and hepatic impairment.

Research Objectives

The pandemic disease COVID-19 is particularly of major importance in Egypt where a heavy population lives. There is an acute need for comprehensive, continuous, and cost-effective health care delivery for infected people. Early detection and strategies for prevention of progression of COVID-19 would make a major difference for these patients and would also be economically beneficial for a resource-constrained country.

This research proposal was employed as a practical strategy for providing a suitable drug combination for possible treatment of COVID-19 infected patients. This drug combination may help to prevent the progression of respiratory complications. This can be achieved through different goals as follows:

1. Screening of different drugs related to different pharmacological classes depending on its possible activity against COVID-19 virus.
2. Providing cost-effective and easy-to-implement treatment strategy for infected patients and/or patients with high risk of developing respiratory failure.
3. Finally, this clinical strategy remains an important goal in improving the Egyptian health state which can save people life and save a lot of money.

Scope of Work

The scope of work will be conducted through:

1. Use of new drug combination of Hydroxychloroquine and Nitazoxanide for treatment of COVID-19 infected people. Since the two drugs exhibit different modes of action, it would be of value in containing the viral infection through targeting different sites in the pathophysiology of the disease.
2. Evaluation of the effect of new drug combination on the symptomatic treatment of newly diagnosed COVID-19 patients through a clinical trial designed according to WHO (clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected) interim guidance published at 13 March 2020.
3. Investigating the impact of new drug combination on the prevention of severe compilations such as acute respiratory distress syndrome (ARDS).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cases of COVID-19 (Positive RT-PCR)
* Newly diagnosed symptomatic patients.
* Adults (18-65 Years old)
* Both sexes

Exclusion Criteria:

* Patients with abnormal liver function (ALT, AST), chronic kidney disease or dialysis (CrCl< 30 ml/min)
* Pregnant women or women who are breastfeeding
* Immunocompromised patients taking medication upon screening
* Subjects with comorbid condition like hypertension, cardiovascular disease, diabetes mellites, asthma, COPD, malignancy
* Patients having allergy to Hydroxychloroquine and/or Nitazoxanide
* Patients with contraindication towards the study medication including retinopathy, G6PD deficiency and QT prolongation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with COVID-19-negative PCR | within 10 days to become PCR negative
  PCR analysis of COVID-19 RNA in patients

SECONDARY OUTCOMES:
Number of patients with improved respiratory rate | within 30 days
  improved breaths per minute for the patients
Number of patients with improved PaO2 | within 30 days
  Change in PaO2 in mmHg of the patients
Number of patients with normalized Serum IL6 | within 30 days
  Serum IL6 in pg/mL of the patients
Number of patients with normalized Serum TNFα | within 30 days
  Serum TNFα in pg/mL of the patients
Number of patients with normalized Serum iron | within 30 days
  Serum iron in microgram/dL of the patients
Number of patients with normalized Serum ferritin | within 30 days
  Serum ferritinin microgram/L of the patients
Number of patients with normalized International normalized ratio "INR" for prothrombin time | within 30 days
  International normalized ratio "INR" for prothrombin time of 2
Number of patients with normalized complete blood count "CBC" | within 30 days
  CBC for lymphocyte count in cells/microliter
The Mortality rate among treated patients | within 30 days
  Mortality rate [number of dead patients/total number of treated patients]

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Okasha, MD, PhD, Principal Investigator — Tanta University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Yu P, Zhu J, Zhang Z, Han Y. A Familial Cluster of Infection Associated With the 2019 Novel Coronavirus Indicating Possible Person-to-Person Transmission During the Incubation Period. J Infect Dis. 2020 May 11;221(11):1757-1761. doi: 10.1093/infdis/jiaa077. PMID 32067043
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Biot C, Daher W, Chavain N, Fandeur T, Khalife J, Dive D, De Clercq E. Design and synthesis of hydroxyferroquine derivatives with antimalarial and antiviral activities. J Med Chem. 2006 May 4;49(9):2845-9. doi: 10.1021/jm0601856. PMID 16640347
- [Background] Marmor MF, Kellner U, Lai TY, Melles RB, Mieler WF; American Academy of Ophthalmology. Recommendations on Screening for Chloroquine and Hydroxychloroquine Retinopathy (2016 Revision). Ophthalmology. 2016 Jun;123(6):1386-94. doi: 10.1016/j.ophtha.2016.01.058. Epub 2016 Mar 16. PMID 26992838
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Raoult D, Houpikian P, Tissot Dupont H, Riss JM, Arditi-Djiane J, Brouqui P. Treatment of Q fever endocarditis: comparison of 2 regimens containing doxycycline and ofloxacin or hydroxychloroquine. Arch Intern Med. 1999 Jan 25;159(2):167-73. doi: 10.1001/archinte.159.2.167. PMID 9927100
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Background] Hong SK, Kim HJ, Song CS, Choi IS, Lee JB, Park SY. Nitazoxanide suppresses IL-6 production in LPS-stimulated mouse macrophages and TG-injected mice. Int Immunopharmacol. 2012 May;13(1):23-7. doi: 10.1016/j.intimp.2012.03.002. Epub 2012 Mar 17. PMID 22430099
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Lu H, Stratton CW, Tang YW. Outbreak of pneumonia of unknown etiology in Wuhan, China: The mystery and the miracle. J Med Virol. 2020 Apr;92(4):401-402. doi: 10.1002/jmv.25678. Epub 2020 Feb 12. No abstract available. PMID 31950516